CLINICAL TRIAL: NCT06579755
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled (Older Adults, Aged >60 to 79 Years) and Open-Label (Adults, Aged 45 to 60 Years), Multicenter Trial to Investigate the Safety and Immunogenicity of a Dengue Tetravalent Vaccine (TDV) Administered Subcutaneously to Adults and Older Adults With or Without Comorbidities in Endemic Areas for Dengue
Brief Title: A Study of Dengue Tetravalent Vaccine (TDV) in Adults (Age 45 to 60 and >60 to 79 Years)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DEN-321
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Dengue Fever
Keywords: Vaccination
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Cohort 1 is randomized and double-blinded. Cohort 2 is non-randomized and open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Tetravalent Dengue Vaccine (TDV) 0.5 mL (Experimental): Participants with the age group greater than (>) 60 to 79 years will receive TDV, 0.5 mL subcutaneous (SC) injections, on Day 1 and Day 90.
  Interventions: Biological: TDV
- Cohort 1: Placebo (Placebo Comparator): Participants with the age group >60 to 79 years will receive placebo (normal saline), 0.5 mL SC injections, on Day 1 and Day 90.
  Interventions: Other: Placebo
- Cohort 2: TDV 0.5 mL (Experimental): Participants with the age group 45 to 60 years will receive TDV, 0.5 mL SC injection, on Day 1 and Day 90.
  Interventions: Biological: TDV

INTERVENTIONS:
Biological: TDV — TDV SC injection.
  Other Names: TAK-003
  Arms: Cohort 1: Tetravalent Dengue Vaccine (TDV) 0.5 mL; Cohort 2: TDV 0.5 mL
Other: Placebo — Placebo SC injection.
  Arms: Cohort 1: Placebo

SUMMARY:
Dengue fever is caused by an infection with the dengue virus. Vaccination with Dengue Tetravalent Vaccine (TDV) can help prevent dengue fever. Researchers have seen that dengue fever now also happens more often in elderly persons. The main aim of this study is to learn more about the side effects of TDV in adult (45 - 60 years) and elderly (60 - 79 years) persons and about TDV's ability to create an immune response in adult and elderly persons. Another aim is to learn about the side effects of TDV in adult and elderly persons in endemic countries who have one or more additional medical conditions (called comorbidities) such as diabetes mellitus, hypertension or a chronic kidney condition.

In this study, participants will receive 2 vaccinations with TDV (the second 3 months after the first).

During the study, participants will visit their study clinic 5 times.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is aged 45 to 79 years at the time of entry into the trial.
2. Participant is male or female.
3. Participant is in good health or has a medical diagnosis of one or more of diabetes mellitus, hypertension, or chronic kidney disease (that is, comorbidities) and are medically stable in the opinion of the investigator at the time of entry into the trial, as determined by medical history and targeted physical examination. Medically stable is defined as no change in diagnoses or chronic medications (dose or class) for medical reasons in the 3 months prior to participating in the trial.
4. Participant has signed and dated a written informed consent form and any required privacy authorization prior to the initiation of any trial procedure, and after the nature of the trial has been explained according to local regulatory requirements.
5. Participant can comply with trial procedures and is available for the duration of follow-up.

Exclusion Criteria:

1. Participant has contraindication(s), warning(s), and/or precaution(s) applicable to vaccination with TDV as specified in the Investigator's Brochure and/or approved product label (as applicable) in the participating country.
2. Participant has a known hypersensitivity or allergy to any of the TDV or placebo components (including excipients).
3. Participant has behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, could interfere with the participant's ability to take part in the trial.
4. Participant has a history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (example, Guillain-Barré syndrome).
5. Participant has an illness, or history of any illness that, in the opinion of the investigator, might interfere with the results of the trial or pose additional risk to the participant due to involvement in this trial.
6. Participant has a known or suspected altered immunocompetence, including:

   1. Chronic administration of oral and/or parenteral steroids at doses considered sufficiently immunosuppressive (example, greater than or equal to [>=] 2 milligram per kilogram [mg/kg] body weight prednisone [or equivalent] for >=14 consecutive days, or >=20 milligram per day [mg/day] prednisone [or equivalent] administered for >=14 consecutive days) within 60 days prior to Day 1 (month [M0]) (note: use of corticosteroids by inhaled, intranasal, intra-articular, bursal, tendon injection, or topical routes is allowed).
   2. Receipt of immunoglobulins and/or any blood products within the 3 months prior to Day 1 (M0) or planned administration during the trial.
   3. Receipt of immunostimulants within 60 days prior to Day 1 (M0).
   4. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months prior to Day 1 (M0).
   5. Human Immunodeficiency Virus (HIV) infection or HIV-related disease.
   6. Hepatitis B virus infection.
   7. Hepatitis C virus infection.
   8. Genetic immunodeficiency.
7. Participant has known or suspected abnormalities of splenic or thymic function.
8. Participant has a known bleeding diathesis, or any condition/medication that may be associated with a prolonged bleeding time.
9. Participant has a serious chronic or progressive disease deemed to be preclusive to trial entry, that is, not medically stable according to the judgment of the investigator.
10. Participant has previously received a vaccination against dengue virus (investigational or licensed).
11. Participant had a clinically significant active infection (as assessed by the investigator) or body temperature >38.0 degree Celsius (>100.4 degree Fahrenheit) within 3 days of intended TDV or placebo administration.
12. Participant has used antipyretics and/or analgesic medications within 24 hours prior to vaccination. The reason for their use (prophylaxis vs treatment) must be documented. Trial entry must be delayed to allow for a full 24 hours to have passed since the last use of antipyretics and/or analgesic medications.
13. Participant has a history of substance or alcohol abuse within the past 2 years.
14. Female participants who are pregnant (that is, a positive or indeterminate pregnancy test).
15. Female participants who are breastfeeding.
16. Female participants of childbearing potential who are sexually active and who have not used any of the acceptable contraceptive methods for at least 2 months prior to Day 1 (M0).
17. Female participants of childbearing potential who are sexually active and who refuse to use an acceptable contraceptive method up to 6 weeks post final vaccination on Day 90 (M3). In addition, they must also be advised not to donate ova during this period.
18. Participant has received any of the following:

    1. A licensed vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to TDV or placebo administration on Day 1 (M0). This includes co-administration with routine vaccines.
    2. A coronavirus vaccine within 14 days prior to TDV or placebo administration.
    3. A vaccine authorized for emergency use within 28 days prior to TDV or placebo administration.
19. Participant is scheduled to receive any other vaccine within 28 days after TDV or placebo administration.
20. Participant is participating in any clinical trial with another investigational product 30 days prior to Day 1 (M0) or intending to participate in another clinical trial at any time during the conduct of this trial.
21. Participant has taken part in any clinical trial of a dengue or other flavivirus (example, West Nile virus) candidate vaccine, except if it is known that the participant received placebo in those trials.
22. Participant or their first-degree relatives are involved in the trial conduct.
23. Participant identified as an employee of the investigator or trial center, with direct involvement in the proposed trial or other trials under the direction of that investigator or trial center.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-04-14 (Estimated); Study Completion 2027-04-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local (Injection Site) Adverse Events (AEs) Within 7 Days Post Vaccination at Day 1 | Within 7 days post-vaccination at Day 1
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered an investigational medical product (IMP); it does not necessarily have to have a causal relationship with IMP administration. Solicited local AEs are injection site pain/tenderness, erythema, and swelling at the vaccination site. All solicited AEs at the injection site will be considered related to the study vaccine administration.
Number of Participants with Solicited Local (Injection Site) Adverse Events (AEs) Within 7 Days Post Vaccination at Day 90 | Within 7 days post-vaccination at Day 90
  Solicited local AEs are injection site pain/tenderness, erythema, and swelling at the vaccination site. All solicited AEs at the injection site will be considered related to the study vaccine administration.
Number of Participants with Solicited Systemic AEs Within 14 Days Post Vaccination at Day 1 | Within 14 days post-vaccination at Day 1
  Solicited systemic AEs include fever (body temperature greater than or equal to [>=] 38 degree Celsius [C], asthenia, malaise, headache, and myalgia.
Number of Participants with Solicited Systemic AEs Within 14 Days Post Vaccination at Day 90 | Within 14 days post-vaccination at Day 90
  Solicited systemic AEs include fever (body temperature >= 38 degree (C), asthenia, malaise, headache, and myalgia.
Percentage of Participants with Solicited Local (Injection Site) AEs by Severity Within 7 Days Post Vaccination at Day 1 | Within 7 days post-vaccination at Day 1
  Solicited local AEs are injection site pain/tenderness, erythema, and swelling at the vaccination site. All solicited AEs at the injection site will be considered related to the study vaccine administration. The AEs will be graded by investigator as Grade 0: none, Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants with Solicited Local (Injection Site) AEs by Severity Within 7 Days Post Vaccination at Day 90 | Within 7 days post-vaccination at Day 90
  Solicited local AEs are injection site pain/tenderness, erythema, and swelling at the vaccination site. All solicited AEs at the injection site will be considered related to the study vaccine administration. The AEs will be graded by investigator as Grade 0: none, Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants with Solicited Systemic AEs by Severity Within 14 Days Post Vaccination at Day 1 | Within 14 days post-vaccination at Day 1
  Solicited systemic AEs include fever (body temperature >= 38 degree (C), asthenia, malaise, headache, and myalgia. The AEs will be graded by investigator as Grade 0: none, Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants with Solicited Systemic AEs by Severity Within 14 Days Post Vaccination at Day 90 | Within 14 days post-vaccination at Day 90
  Solicited systemic AEs include fever (body temperature >= 38 degree (C), asthenia, malaise, headache, and myalgia. The AEs will be graded by investigator as Grade 0: none, Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants with Any Unsolicited AEs Within 28 Days Post Vaccination at Day 1 | Within 28 days post-vaccination at Day 1
  An unsolicited AE is any AE reported by the participant that is not specified as a solicited AE or is specified as a solicited AE but starts outside the period for reporting a solicited AE (that is, 7 days and 14 days in total including the day IMP administration).
Percentage of Participants with Any Unsolicited AEs Within 28 Days Post Vaccination at Day 90 | Within 28 days post-vaccination at Day 90
  An unsolicited AE is any AE reported by the participant that is not specified as a solicited AE or is specified as a solicited AE but starts outside the period for reporting a solicited AE (that is, 7 days and 14 days in total including the day of IMP administration).
Percentage of Participants with a Serious Adverse Event (SAE) | From first vaccination on Day 1 through the end of trial (up to Day 270)
  An SAE is defined as any untoward medical occurrence that: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/ incapacity, leads to a congenital anomaly/birth defect in the offspring of a participant, is an important medical event.
Geometric Mean Titers (GMTs) of Neutralizing Antibodies by Microneutralization Test (MNT) for Each of the 4 Dengue Virus Serotypes at Day 120 | At Day 120
  GMTs of neutralizing antibodies will be measured by microneutralization test 50% [MNT50] for each of the 4 Dengue Serotypes in all participants. The 4 dengue virus serotypes are dengue virus (DENV)-1, DENV-2, DENV-3 and DENV-4.

SECONDARY OUTCOMES:
Number of Participants with Solicited Local (Injection Site) AEs Within 7 Days Post Vaccination at Day 1 and Day 90 (With Comorbidities) | Within 7 days post-vaccination at Day 1 and Day 90
  Solicited local AEs are injection site pain/tenderness, erythema, and swelling at the vaccination site. All solicited AEs at the injection site will be considered related to the study vaccine administration.
Number of Participants with Solicited Systemic AEs Within 14 Days Post Vaccination at Day 1 and Day 90 (With Comorbidities) | Within 14 days post-vaccination at Day 1 and Day 90
  Solicited systemic AEs include fever (body temperature >= 38 degree (C), asthenia, malaise, headache, and myalgia.
Percentage of Participants with Solicited Local (Injection Site) AEs by Severity Within 7 days Post Vaccination at Day 1 and Day 90 (With Comorbidities) | Within 7 days post-vaccination at Day 1 and Day 90
  Solicited local AEs are injection site pain/tenderness, erythema, and swelling at the vaccination site. All solicited AEs at the injection site will be considered related to the study vaccine administration. The AEs will be graded by investigator as Grade 0: none, Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants with Solicited Systemic AEs by Severity (With Comorbidities) | Within 14 days post-vaccination at Day 1 and Day 90
  Solicited systemic AEs include fever (body temperature >= 38 degree (C), asthenia, malaise, headache, and myalgia. The AEs will be graded by investigator as Grade 0: none, Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants with Any Unsolicited AEs Within 28 Days Post Vaccination (With Comorbidities) | Within 28 days post-vaccination at Day 1 and Day 90
  An unsolicited AE is any AE reported by the participant that is not specified as a solicited AE or is specified as a solicited AE but starts outside the period for reporting a solicited AE (that is, 7 days and 14 days in total including the day IMP administration).
Percentage of Participants with a SAE (With Comorbidities) | From first vaccination on Day 1 through the end of trial (up to Day 270)
  An SAE is defined as any untoward medical occurrence that: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/ incapacity, leads to a congenital anomaly/birth defect in the offspring of a participant, is an important medical event.
Geometric Mean Titers by MNT for Each of the 4 Dengue Virus Serotypes | Day 1, Day 30, Day 90 and Day 270
  GMTs of neutralizing antibodies will be measured by MNT50 for each of the 4 dengue serotypes in all participants. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Geometric Mean Titers by MNT for Each of the 4 Dengue Virus Serotypes (With Comorbidities) | Day 1, Day 30, Day 90, Day 120 and Day 270
  GMTs of neutralizing antibodies will be measured by MNT50 for each of the 4 dengue serotypes. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Seropositivity Rate for Each of the 4 Dengue Virus Serotypes | Day 1, Day 30, Day 90, Day 120 and Day 270
  Seropositivity rate is defined as the percentage of participants with MNT titer >=10 against each of the four dengue virus serotypes in all participants. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Seropositivity Rate for Each of the 4 Dengue Virus Serotypes (With Comorbidities) | Day 1, Day 30, Day 90, Day 120 and Day 270
  Seropositivity rate is defined as the percentage of participants with MNT titer >=10 against each of the four dengue virus serotypes. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Seropositivity Rate for Multiple (2, 3, or 4) Dengue Virus Serotypes | Day 1, Day 30, Day 90, Day 120 and Day 270
  Seropositivity rate is defined as the percentage of participants with MNT titer >=10 against multiple (2, 3, or 4) dengue virus serotypes in all participants. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Seropositivity Rate for Multiple (2, 3, or 4) Dengue Virus Serotypes (With Comorbidities) | Day 1, Day 30, Day 90, Day 120 and Day 270
  Seropositivity rate is defined as the percentage of participants with MNT titer >=10 against multiple (2, 3, or 4) dengue virus serotypes. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (7):
- Fundacion Huesped - PPDS, Buenos Aires, Argentina
- Brazil (2):
  - Associacao Obras Sociais Irma Dulce Hospital Santo Antonio, Salvador, Estado de Bahia
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto Hospital de Base - PPDS, São José do Rio Preto, São Paulo
- Singapore (2):
  - Singapore General Hospital (SGH), Singapore
  - Tan Tock Seng Hospital, Singapore
- Thailand (2):
  - Ramathibodi Hospital, Ratchathewi, Bangkok
  - Hospital for Tropical Diseases, Ratchathewi, Krung Thep Maha Nakhon-Bangkok

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/38711336188b488b??page=1&idFilter=DEN-321